CLINICAL TRIAL: NCT03945110
Title: Intravesical Glycosaminoglycan Instillation Following Spinal Cord Injury and Early Urinary Tract Infections; Safety and Feasibility Study
Brief Title: Intravesical Glycosaminoglycan Instillation and Urinary Tract Infection in Acute Spinal Cord Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Western Australia (Other)
Collaborators: Royal Perth Hospital (Other); Fiona Stanley Hospital (Other); Perth Urology Clinic (Unknown)
Responsible Party: Principal Investigator, Sarah Dunlop, Coordinating Principal Investigator, The University of Western Australia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RA/4/20/5351
Record Dates: First submitted 2019-05-03; First posted 2019-05-10 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Consenting participants meeting eligibility criteria will join the intervention arm of trial; participants not meeting eligibility criteria and/or unwilling to receive intervention but consenting for data collection on bladder health measures for the study duration will join the non-intervention (standard care only) arm of trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Patients in this Arm will receive a series of seven iAluRil® intravesical instillations over a 12-week period as follows: Once per week for 4 weeks; then once every two weeks for 4 weeks; then once 4 weeks later.
  Interventions: Device: iAluRil® intravesical instillations
- Arm B (No Intervention): Patients in this Arm will receive usual bladder care only.
- Arm C (Experimental): Patients in this Arm will be Spinal Urology Outpatients or Inpatients who are eligible for inclusion and experiencing significant urinary tract infection recurrence and/or complications. Patients will receive a series of seven iAluRil® intravesical instillations over a 12-week period as follows: Once per week for 4 weeks; then once every two weeks for 4 weeks; then once 4 weeks later. Patients will be encouraged and supervised to self-administer iAluRil® intravesical instillations.
  Interventions: Device: iAluRil® intravesical instillations

INTERVENTIONS:
Device: iAluRil® intravesical instillations — 50ml of a sterile solution of sodium hyaluronate (1.6% 800mg/50ml) and sodium chondroitin sulphate (2% - 1 g/50ml) is administered intravesically (directly into the bladder) via a pre-filled syringe connected to a catheter and held in the bladder for at least 30 minutes.
  Other Names: Intravesical glycosaminoglycan (GAG) therapy
  Arms: Arm A; Arm C

SUMMARY:
The purpose of this study is to assess the safety and feasibility of administering glycosaminoglycan (GAG) therapy, iAluRil®, intravesically in individuals with acute spinal cord injury (SCI), commencing within the first ten days of injury, to prevent early urinary tract infections.

DETAILED DESCRIPTION:
iAluRil®, listed as a medical device on the Australian Therapeutic Goods Registry (ATGR), contains both hyaluronic acid and chondroitin sulphate. This trial utilises iAluRil® for the same clinical indication as it is listed for on the ATGR, i.e. to re-establish the glycosaminoglycan (GAG) layers of the urothelial vesical tissue in cases in which their loss can cause problems, such as recurrent urinary tract infection in neurologically intact populations, but in a specific and vulnerable patient population (acute SCI). The trial will demonstrate the safety and feasibility of providing a series of iAluRil® treatments in early acute SCI, and provide an indication of effectiveness to prevent early urinary tract infections (compared to current standard infection control), informing researchers about the suitability of conducting a large randomised controlled clinical trial with this intervention.

An 'Intervention post-UTI' arm for eligible inpatients and outpatients with SCI who have significant recurrent UTIs, will allow equivalent data collection and observations, informing researchers about a trial to reduce UTI recurrence during sub-acute/chronic SCI. Additionally, these patients will self-administer iAluRil® treatments providing data on the feasibility of SCI patients self-administering iAluRil® treatments.

ELIGIBILITY:
Arm A & B Inclusion Criteria:

- Patients hospitalised at Royal Perth Hospital (RPH) in Western Australia following first acute traumatic SCI (with any degree of neurological impairment)

Arm A & B Exclusion Criteria:

* Admitted to a hospital outside of Western Australia following SCI (prior to RPH)
* Unable to commence intervention within 10 days post-SCI
* Bladder or urethral trauma on admission
* Known history of bladder cancer or other bladder pathology
* Known hypersensitivity to hyaluronic acid, sodium salt or sodium chondroitin sulphate
* Diagnosis of a symptomatic urinary tract infection prior to commencing treatment
* Pregnancy
* Previous neurological disorder
* Inability to provide own consent due to intellectual, mental or cognitive impairment

Arm C Inclusion Criteria:

* Previous traumatic or non-traumatic (sudden onset) SCI
* Experience significant, recurrent UTIs (in the opinion of the treating Spinal / Urology Consultant
* Willing and able to partake in all study requirements
* Emptying bladder via intermittent catheterisation (self or carer administered)

Arm C Exclusion Criteria:

* Bladder or urethral trauma
* Known history of bladder cancer or other bladder pathology
* Known hypersensitivity to hyaluronic acid sodium salt or sodium chondroitin sulphate
* Pregnancy
* Previous neurological disorder
* Inability to provide own consent due to intellectual, mental or cognitive impairment
* Significant known history of Autonomic Dysreflexia associated with urological procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Proportion of eligible traumatic SCI patients who start iAluRil within 10 days post injury | 10 days pos-SCI for each participant
  The proportion of eligible traumatic SCI patients who were urinary tract infection (UTI) free, able to provide informed consent and receive the first iAluRil instillation within 10 days of SCI

SECONDARY OUTCOMES:
Proportion of eligible traumatic SCI patients administered iAluRil within 10 days of SCI who completed seven iAluRil instillations as per protocol over 12 weeks | 12 weeks (+/- 1 week) following recruitment for each participant
  The proportion of eligible traumatic SCI patients administered iAluRil within 10 days who then completed seven iAluRil instillations as per protocol over 12 weeks
Median time to first symptomatic UTI | Date of SCI to date of hospital discharge, an average of three months
  Median time (days) between SCI and first medically diagnosed symptomatic UTI
Incidence of symptomatic UTI/100 patient days | Date of SCI to date of hospital discharge, an average of three months
  Number of medically diagnosed symptomatic UTIs per 100 days of hospitalisation
Incidence of other urological complications/100 patient days | Date of SCI to date of hospital discharge, an average of three months
  Number of other (non-UTI) urological complications per 100 days of hospitalisation
Length of hospital stay | Date of SCI to date of hospital discharge, an average of three months
  Number of days of initial hospitalisation (acute and subacute/rehabilitation)
Bladder-related quality of life - bladder management difficulties | Conducted at 12 weeks post recruitment and at 24 weeks post recruitment for each participant
  Validated SCI-QOL Questionnaire: 'Bladder Management Difficulties SF8a'
Bladder-related quality of life - bladder complications | Conducted at 12 weeks post recruitment and at 24 weeks post recruitment for each participant
  Validated SCI-QOL Questionnaire: 'Bladder Complications'
Incidence of Adverse Events | During 12-week intervention period for each participant
  Incidence of significant adverse events requiring medical intervention and/or impacting on hospital length of stay in Arm A will be described

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Dunlop, PhD, Principal Investigator — The University of Western Australia
Locations (1):
- Royal Perth Hospital, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for primary and secondary outcomes that form the basis of the final scientific paper will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available upon request immediately following publication and indefinitely thereafter via a link to the relevant section of The University of Western Australia's research repository.
Access Criteria: Data will be available upon request to Researchers providing a methodologically sound research proposal, for the purpose of achieving the aims in this proposal. Proposals should be directed to sarah.dunlop@uwa.edu.au

REFERENCES:
- [Background] Damiano R, Cicione A. The role of sodium hyaluronate and sodium chondroitin sulphate in the management of bladder disease. Ther Adv Urol. 2011 Oct;3(5):223-32. doi: 10.1177/1756287211418723. PMID 22046200
- [Background] Manas A, Glaria L, Pena C, Sotoca A, Lanzos E, Fernandez C, Riviere M. Prevention of urinary tract infections in palliative radiation for vertebral metastasis and spinal compression: a pilot study in 71 patients. Int J Radiat Oncol Biol Phys. 2006 Mar 1;64(3):935-40. doi: 10.1016/j.ijrobp.2005.09.016. Epub 2006 Jan 10. PMID 16376493
- [Background] Damiano R, Quarto G, Bava I, Ucciero G, De Domenico R, Palumbo MI, Autorino R. Prevention of recurrent urinary tract infections by intravesical administration of hyaluronic acid and chondroitin sulphate: a placebo-controlled randomised trial. Eur Urol. 2011 Apr;59(4):645-51. doi: 10.1016/j.eururo.2010.12.039. Epub 2011 Jan 18. PMID 21272992
- [Derived] King GK, Goodes LM, Hartshorn C, Thavaseelan J, Jonescu S, Watts A, Rawlins M, Woodland P, Synnott EL, Barrett T, Hayne D, Boan P, Dunlop SA. Intravesical hyaluronic acid with chondroitin sulphate to prevent urinary tract infection after spinal cord injury. J Spinal Cord Med. 2023 Sep;46(5):830-836. doi: 10.1080/10790268.2022.2089816. Epub 2022 Jul 6. PMID 35792831